CLINICAL TRIAL: NCT03881878
Title: Docetaxel Plus Atezolizumab Plus Herceptin SC and Pertuzumab (TAHP) for Patients With HER2-positive Early Breast Cancer and Subsequent Atezolizumab Plus Herceptin SC and Pertuzumab (AHP) Adjuvant tHerapy After Surgery
Brief Title: TAHP for Patients With HER2-positive Early Breast Cancer and Subsequent AHP Adjuvant tHerapy After Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Clinical Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01-064
Record Dates: First submitted 2019-03-11; First posted 2019-03-20 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Intervention Model Description: (A, Neoadjuvant setting): TAHP (Docetaxel, Atezolizumab, Trastuzumab sc and Pertuzumab) D1 X 6 cycles q3weeks, intravenous(IV) administration
  (B, Adjuvant setting) : patients with pCR: AHP(Atezolizumab, Trastuzumab sc and Pertuzumab) D1 X 11-12 cycles q3weeks
  patients with non-pCR: Doxorubicin plus cyclophosphamide: D1 X 4cycles q3weeks followed by AHP (Atezolizumab, Trastuzumab sc and Pertuzumab) D1 X 11-12 cycles q3weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pathologic Complete response (Experimental): (A, Neoadjuvant setting): D1 X 6 cycles, q3weeks
  * Docetaxel (75mg/m2, IV)
  * Atezolizumab (1200mg, IV)
  * Trastuzumab (600mg, SC)
  * Pertuzumab (840mg loading dose at Cycle 1 followed by 420mg, IV)
  (B, Adjuvant setting) : D1 X 11-12 cycles, q3weeks
  * Atezolizumab (1200mg, IV)
  * Trastuzumab (600mg, SC)
  * Pertuzumab (420mg, IV)
  Interventions: Drug: TAHP and AHP
- non-pathologic Complete response (Experimental): (A, Neoadjuvant setting): D1 X 6 cycles, q3weeks
  * Docetaxel (75mg/m2, IV)
  * Atezolizumab (1200mg, IV)
  * Trastuzumab (600mg, SC)
  * Pertuzumab (840mg loading dose at Cycle 1 followed by 420mg, IV)
  (B, Adjuvant setting) :
  * Doxorubicin(60mg/m2) plus cyclophosphamide (600mg/m2) : D1 X 4cycles q3weeks followed by
  * Atezolizumab (1200mg, IV), Trastuzumab (600mg, SC) and Pertuzumab (420mg, IV) D1 X 11-12 cycles q3weeks
  Interventions: Drug: TAHP plus AC and AHP

INTERVENTIONS:
Drug: TAHP and AHP — (A, Neoadjuvant setting): D1 X 6 cycles, q3weeks
  * Docetaxel (75mg/m2, IV)
  * Atezolizumab (1200mg, IV)
  * Tastuzumab (600mg, SC)
  * Pertuzumab (840mg loading dose at Cycle 1 followed by 420mg, IV)
  (B, Adjuvant setting) : patients with pCR:D1 X 11-12 cycles, q3weeks
  * Atezolizumab (1200mg, IV)
  * Trastuzumab (600mg, SC)
  * Pertuzumab (420mg, IV)
  Arms: pathologic Complete response
Drug: TAHP plus AC and AHP — (A, Neoadjuvant setting): D1 X 6 cycles, q3weeks
  * Docetaxel (75mg/m2, IV)
  * Atezolizumab (1200mg, IV)
  * Tastuzumab (600mg, SC)
  * Pertuzumab (840mg loading dose at Cycle 1 followed by 420mg, IV)
  (B, Adjuvant setting) : patients with non-pCR
  * Doxorubicin(60mg/m2) plus cyclophosphamide (600mg/m2) D1 X 4cycles q3weeks followed by
  * Atezolizumab (1200mg, IV), Trastuzumab (600mg, SC) and Pertuzumab (420mg, IV) D1 X 11-12 cycles q3weeks
  Arms: non-pathologic Complete response

SUMMARY:
This study was phase IB-II clinical trial that designed to evaluate the efficacy and safety of docetaxel + atezolizumab + Herceptin sc plus pertuzumab(TAHP) plus adjuvant therapy of atezolizumab + trastuzumab + pertuzumab(AHP) after surgery in female patients with HER2-positive early breast cancer.

Adjuvant AHP (atezolizumab + Herceptin SC + pertuzumab) will be continued for remaining 1 year.

For non-p CR patients, they are going to treat with 4 cycles of AC rather than Taxane only before AHP adjuvant therapy.

DETAILED DESCRIPTION:
A, Neoadjuvant setting); 6 cycles q3weeks, intravenous(IV) administration

* Docetaxel (75mg/m2, intravenous(IV)) Day(D)1
* Atezolizumab (1200mg, IV) D1
* Herceptin sc (600mg subcutaneous(SC))D1
* Pertuzumab (840mg loading dose at Cycle 1 followed by 420mg(IV))D1

B, Adjuvant setting : 11-12 cycles q3weeks [patients with pCR]

* Atezolizumab (1200mg, IV)
* Trastuzumab (600mg, SC)
* Pertuzumab (420mg, IV) D1

[patients with non-pCR]

* Doxorubicin(60mg/m2), cyclophosphamide (600mg/m2) D1 X 4cycles 3weeks
* Atezolizumab (1200mg, IV)
* Trastuzumab (600mg, SC)
* Pertuzumab (420mg, IV) D1 X 11-12 cycles q3weeks

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult, female ≥ 18 years old at the time of informed consent
2. Patient has histologically confirmed diagnosis of breast cancer
3. Patients with locally advanced breast cancer (T2-3N0-3)
4. Patients with early breast cancer with high-risk (T1cN1)
5. Patients with locally advanced inflammatory breast cancer
6. Patient has HER2-positive breast cancer as 3+ by IHC or in-situ hybridization (ISH) amplified BC patients
7. ER+ or ER-
8. Agree to informed consent and willing and able to comply with the protocol
9. Available pre-chemotherapy and surgery tissue (except pCR)
10. For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study drugs. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

    Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.
11. Patient has adequate bone marrow and organ function
12. LVEF ≥55% at baseline

Exclusion Criteria:

1. HER2-negative in surgery sample
2. Tumor size less than 2cm or and N0
3. Patients who have metastatic disease (M1)
4. Patients who are not available tumor tissue
5. Pregnant or lactating or intending to become pregnant during or within 7 months after the last dose of study treatment
6. Patients who have serious underlying co-morbidities which could cause end-organ dysfunction
7. Any previous treatment against including chemo, hormonal therapy
8. Administration of a live, attenuated vaccine within 4 weeks before Day 1 or anticipation that such a live attenuated vaccine will be required during the study
9. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
10. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
11. Patients with prior allogeneic stem cell or solid organ transplantation
12. History of autoimmune disease including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
13. History of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) or evidence of active pneumonitis on screening chest computed tomography scan
14. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
15. History of HIV infection, active hepatitis B (chronic or acute), or hepatitis C infection. Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [anti-HBc] test) are eligible.
16. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction assay (PCR) is negative for HCV RNA
17. Active tuberculosis
18. Severe infections within 4 weeks prior to Day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. Signs or symptoms of significant infection within 2 weeks prior to Day 1
19. Received oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
20. Previous or concomitant malignancy of any other type that could affect compliance with the protocol or interpretation of results. Patients with curatively treated basal cell carcinoma of the skin or in situ cervix cancer are generally eligible
21. Congestive heart failure or abnormal LVEF(LVEF is not ≥55% at baseline)
22. Total bili >1.5 ULN (except for Gilbert's syndrome), AST/ALT > 1.5 ULN, ALP > 2.5 ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2019-05-27 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic CR(pCR) rate of neo-adjuvant chemotherapy | Pathologic Clinical response is perforemed after end of cycle 6 (each cycle is 21days).
  pCR rate of neoadjuvant chemotherapy with the patients with HER2+ EBC

SECONDARY OUTCOMES:
Event free survival(EFS) | 3 years
  Event free survival of the patient with pCR vs. non-pCR

OTHER OUTCOMES:
Adverse events will be measured by the CTCAE scale, version 5.0 | 1 year
  safety and toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ahn HK, Sim SH, Suh KJ, Kim MH, Jeong JH, Kim JY, Lee DW, Ahn JH, Chae H, Lee KH, Kim JH, Lee KS, Sohn JH, Choi YL, Im SA, Jung KH, Park YH. Response Rate and Safety of a Neoadjuvant Pertuzumab, Atezolizumab, Docetaxel, and Trastuzumab Regimen for Patients With ERBB2-Positive Stage II/III Breast Cancer: The Neo-PATH Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2022 Sep 1;8(9):1271-1277. doi: 10.1001/jamaoncol.2022.2310. PMID 35797012